CLINICAL TRIAL: NCT02379936
Title: Evaluation of a Point of Care Analyzer for Lactate Dehydrogenase, HildaNeo, as Support for Decisions When Admitting Newborn to the Neonatal Wards at NPH
Brief Title: Evaluation of Lactate Dehydrogenase as Decision Support for Admissions to Neonatal Ward
Acronym: HildaNeoHan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Children's Hospital, Vietnam (Other)
Collaborators: Calmark Sweden AB (Unknown); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Khu Khanh Thi, Dung, Vice director NPH; Assoc Prof., MD, PhD, National Children's Hospital, Vietnam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HildaNeo test study Vietnam
Record Dates: First submitted 2013-08-20; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-02

CONDITIONS: Neonatal; Asphyxia
Keywords: Classification; HIE; Infections; Lactate dehydrogenase; Intensive Care
MeSH Terms: conditions — Asphyxia; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The NeoHilda Point of care method (Active Comparator): Evaluating baby including lactate dehydrogenase Levels measured in umbilical core blood using the fast point of care method called Neo Hilda
  Interventions: Device: The Neo Hilda; Device: iPhone 4S
- No Measurement of LDH (Sham Comparator): Evaluating baby without Lactate dehydrogenase result
  Interventions: Procedure: Traditional evaluation

INTERVENTIONS:
Device: The Neo Hilda — This is a procedure that measures Lactate dehydrogenase in a fast and reliable way from only 10 microliter of blood. Using a small point of care card and a Smartphone for analysis.
  Point of care method
  Other Names: Neo Hilda, Calmark Sweden AB
  Arms: The NeoHilda Point of care method
Procedure: Traditional evaluation — Traditional way of evaluation
  Arms: No Measurement of LDH
Device: iPhone 4S
  Arms: The NeoHilda Point of care method

SUMMARY:
The immediate newborn period is the period of highest morbidity in life. Early signs of serious disease are often vague and difficult to interpret for the non- specialist. Screening lists of clinical signs are useful but have unsatisfactory specificity or sensitivity, cover only one or two diseases, and are complicated to handle in low resource settings.

In critically ill newborns, organ failure to one or multiple organ systems is frequently seen due to inadequate circulation to the tissues. Critical disease will cause hypoxia ischemia of the cells in the affected organs followed by energy deficiency. Independently of the condition causing the energy deficiency this will start a series of events, which initially cause a leaking cell membrane leading to that intracellular components, i.e. the enzyme Lactate dehydrogenase (LDH), will leak out into the blood. Previous research in newborns suggests that LDH is a clinically interesting early predictor of serious illness and may thus serve as an important complement to the clinical examination. If the LDH level is elevated the health care personnel will realize that something is wrong and call for appropriate measures.

Today LDH analysis is performed at the Dept. of Clinical Chemistry with an inexpensive and accurate method. However, this method needs relatively large blood volumes and the delay between blood sampling and results is rather long, often several hours. In addition LDH is sensitive to hemolysis, which is quite common in blood sampling in newborns. When this is detected at the laboratory a new sample will be needed, thus delaying the result even more. Also, smaller health care facilities rarely have the laboratory equipment needed for the analysis of LDH.

The Swedish company Calmark Sweden AB is now launching a point-of-care technology for LDH analysis called "Hilda Neo". LDH is analyzed on an easy-to-use consumable test card together with an "App" on an ordinary smartphone (in the planned study, iPhone 4S). The result is presented within minutes and presence of hemolysis will be simultaneously detected on the device.

The investigators speculate that the use of such a LDH test could serve as a diagnostic help for health-care staff in Vietnam in making the decision when to send a potentially sick newborn to a higher level neonatal unit (in this case the NICU at NPH, Hanoi)

DETAILED DESCRIPTION:
Patients and Methods At admission to NPH, newborn (GA >32 w, ≤36h old) infants referred to NPH with suspect or probable clinical signs of illness for which the physician on call considers that a blood sample is needed will be included in the study when a doctor taking part in the study is present at the ward. When a blood test is indicated, around 2 ml of blood is routinely drawn including an extra 0.1 ml blood for analysis of LDH using the Hilda Neo card.

When an infant fulfils the inclusion criteria the physician on duty will open a downloaded "App" on the provided smartphone and take a photo of the first page of the study protocol including the patients study number time of birth, and the result of the clinical investigation on a simple clinical score protocol. Then the physician presses a "randomise button" on the smartphone to randomise to using the Hilda Neo card or to routine care. If randomised to the Hilda Neo card use the "app" gives instructions how to use the card and guides through the different steps of the test. The result of the LDH test will be presented to the physician immediately at the point-of-care and can be used in the clinical decisions.

To prepare for a following study of the usefulness of LDH when deciding if a baby is ready for transfer from the NICU to ordinary care all included infants will have an LDH test at the routine clinical laboratory daily when other blood samples are drawn. The investigators believe that two LDH tests at 6 - 24 hour intervals are needed for that question. The reason for using two tests with an interval is that a high single LDH value can be expected in a large number of the infants because of the preceding disease while a decreasing value might be a better predictor of an improving status.

An evaluation protocol is filled in by the neonatologist in the ward 80-96h after admission or, if earlier, at discharge or death. The classification of the protocols into "need for" and "no need for intensive care resources" will be done independently by two senior neonatologists, both blinded to the LDH results from the Hilda card and the routine clinical laboratory.

The outcome that will be reported is the number of patients admitted to correct level of care, NICU or level 2 unit, in the two groups the admitting doctor has or has not access to plasma LDH respectively.

The definitions of correct or not correct admission level were:

1. Admitted to NICU care: correct decision=The patient did fulfil the criteria for referral to NICU during the first 80 and 96h after admission.
2. Admitted to NICU care: not correct decision=The patient did not fulfil the criteria for referral to NICU during the first 80 to 96h after admission.
3. Admitted to level 2 unit: correct decision=The patient did not fulfil the criteria for referral to NICU during the first 80 to 96h after admission.
4. Admitted to level 2 unit: not correct decision= The patient did fulfil the criteria for referral to NICU between 80 and 96h after admission The classification of the protocols into "fulfil or not fulfil the criteria for intensive care resources" was done independently by two senior neonatologists, both blinded to the LDH results from the Hilda card and the routine clinical laboratory.

The criteria for "fulfil the criteria for intensive care resources" were that shock-, ventilator-, CPAP- treatment, blood exchange, parenteral nutrition or other procedures demanding NICU capacity in the actual setting were performed during the first 80 - 96 hours after admission.

For calculation of the number of patients needed for the study outcome "right decision" in relation to "wrong decision" will be used, see below under Power.

The results will be recorded on the paper protocol forms, which are kept with the clinical record of the patient. The results will also be kept as a photo using the Smart phone App where it can be read only until the picture has been sent to the register. When the picture comes to the register it is identified only by its study number. Name and identity together with the study number is taken from the patient record to a separate register, which is securely kept by one authorized person in order for future supplementary information. The data recorded for the study are those normally recorded for a NICU patient and the doctors evaluation of the Hilda card.

The de-identified protocols will be saved, processed and analysed with the statistical program SPSS. Only persons involved in the study will have access to the data registered.

Based on going (Itzel et.al) and previously conducted research a LDH activity exceeding 600U/L will be considered as increased.

Power calculation In the investigators earlier study about 75% of the babies admitted to the NICU did not need intensive care procedures during the first week. To detect a reduction from 75 to 50% according to outcome above would need 58 patients in the test and the control group respectively. The control group here is the group that is not admitted to the NICU ward but to the ordinary care ward.

If there are technical or other problems with the Hilda Neo test that might influence the primary outcome the study will include 58 babies after the problem has been solved.

The background factors and the criteria for need of intensive care that will be noted are presented on the protocols, (n= 120+20 patients)

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to the neonatal ward above 32w of age, considered for blood sampling.

Exclusion Criteria:

* Parental consent missing
* Gestational age less than 33 weeks postnatal age above 36 hours

Ages: 2 Minutes to 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The number of patients admitted to correct level of care, NICU or level 2 unit, in the two groups the admitting doctor has or has not access to plasma LDH respectively. | at 96 hours after admission
  The definitions of correct or not correct admission level were:
  1. Admitted to NICU care: correct decision=The patient did fulfil the criteria for referral to NICU during the first 80 and 96 hours after admission.
  2. Admitted to NICU care: not correct decision=The patient did not fulfil the criteria for referral to NICU during the first 80 to 96 hours after admission.
  3. Admitted to level 2 unit: correct decision=The patient did not fulfil the criteria for referral to NICU during the first 80 to 96 hours after admission.
  4. Admitted to level 2 unit: not correct decision= The patient did fulfil the criteria for referral to NICU between 80 and 96 hours after admission

SECONDARY OUTCOMES:
The proportion of admitted infants diagnosed as HIE had an LDH value according to the Hilda Card over cut off 600 U/l. | 30 days after completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Khu TK Dung, Ass prof., Principal Investigator — National Hospital of Pediatrics; Birger Winbladh, Professor, Study Director — Karolinska Institutet
Locations (1):
- Neonatal unit, National hospital of Pedriatrics, Hanoi, Hanoi, Vietnam

REFERENCES:
- [Background] Karlsson M, Dung KT, Thi TL, Borgstrom E, Jonstam K, Kasstrom L, Winbladh B. Lactate dehydrogenase as an indicator of severe illness in neonatal intensive care patients: a longitudinal cohort study. Acta Paediatr. 2012 Dec;101(12):1225-31. doi: 10.1111/apa.12014. PMID 22963670
- [Background] Karlsson M, Wiberg-Itzel E, Chakkarapani E, Blennow M, Winbladh B, Thoresen M. Lactate dehydrogenase predicts hypoxic ischaemic encephalopathy in newborn infants: a preliminary study. Acta Paediatr. 2010 Aug;99(8):1139-44. doi: 10.1111/j.1651-2227.2010.01802.x. Epub 2010 Mar 19. PMID 20236255
- [Background] Wiberg-Itzel E, Akerud H, Andolf E, Hellstrom-Westas L, Winbladh B, Wennerholm UB. Association between adverse neonatal outcome and lactate concentration in amniotic fluid. Obstet Gynecol. 2011 Jul;118(1):135-142. doi: 10.1097/AOG.0b013e318220c0d4. PMID 21691171
- [Background] Thoresen M, Liu X, Jary S, Brown E, Sabir H, Stone J, Cowan F, Karlsson M. Lactate dehydrogenase in hypothermia-treated newborn infants with hypoxic-ischaemic encephalopathy. Acta Paediatr. 2012 Oct;101(10):1038-44. doi: 10.1111/j.1651-2227.2012.02778.x. Epub 2012 Jul 27. PMID 22775455